CLINICAL TRIAL: NCT07064941
Title: Effect of Aerobic Exercise Paired With Strength Conditioning on Bone Health in Patients With Thalassemia
Brief Title: Effect of Exercise on Body Composition and Bone Health in Patients With Thalassemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thal Exercise
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Thalassemia
Keywords: Exercise; Body composition; Bone; Muscle function
MeSH Terms: conditions — Thalassemia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a delayed start interventional study where subjects serve as their own controls. Each subject will first participate in a 12 week usual care period in which they will not change their activity, followed by a 12 week exercise intervention (Period 1) and end with an additional 24 weeks of the exercise intervention (Period 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual Activity (Other): Subjects will participate in usual daily activities during this period
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise for 30 min a day 5x a week with a choice between Aerobic or strength training. Subjects will choose an aerobic activity to perform 3x/week (e.g. brisk walking, hiking, jogging). They will start at 15-20 min/day depending on fitness level and build up by 5 min intervals/week as tolerated to 50 min/day or 150 min/week by 12 weeks. Subjects will choose strength exercises to perform 2x/week, on days separate from aerobic activity. They will start with 1-2 exercises (e.g. squats, lunges, planks with and without resistance) and gradually add exercises to include all muscle groups (arms, legs, chest, back, abdomen). Start with 2 sets of 10 reps, and work up to 3 sets of 15 reps of given exercises.

SUMMARY:
The goal of this clinical trial is to determine if a weight bearing exercise intervention can improve body composition and bone health in adolescents and adults with Thalassemia.

The main questions it aims to answer are:

* Does participation in a 12-week weight bearing exercise intervention change total body lean mass and percentage body fat (as assessed by DXA) in adolescents and adults with Thalassemia?
* Does participation in a 12-week weight bearing exercise intervention change muscle function (assessed by hand grip strength, sit to stand and vertical jump) and endurance (assessed by the 6 minute walk test) in adolescents and adults with Thalassemia?
* Does participation in a 36 week weight bearing exercise intervention (30 min/day; 5x/week) change bone mineral density as assessed by DXA in adolescents and adults with Thalassemia?

Researchers will compare participants' change in body composition, muscle mass, and muscle function during a "Usual Activity" period (12 weeks) with an exercise intervention (Period 1: 12 weeks) to see if exercise can improve body composition and muscle function.

The intervention will then be extended an additional 24 weeks for a total of 36 weeks of exercise (Period 2) to explore the change in bone mineral density between between "Usual Activity" and "Exercise Intervention" (Period 2) in individuals with Thalassemia.

During the intervention period, participants will engage in a self-directed exercise regime of either weight bearing aerobic exercise or strength training exercises (30 min/day; 5x/week).

ELIGIBILITY:
Inclusion Criteria:

* Age: 14 - 40 years
* BMD Z-score at any skeletal site < -1.0
* Diagnosed with thalassemia (any genotype, regardless of transfusion dependency)
* Vitamin D (25-Hydroxy) drawn within the previous 12 months >20 ng/mL
* English speaking, able to consent

Exclusion Criteria:

* Patients who self-identify as 'exercisers' e.g. routinely exercise for minimum of 45 min/day, 5x/week
* Pregnant (unable to conduct bone density measurements in pregnant females)
* Hypogonadal, must be on replacement sex hormone therapy for min of 6 months
* Cardiac T2* by Magnetic Resonance Imaging of <20 ms (e.g. evidence of cardiac iron overload)
* Recent long bone or vertebral fracture (within the last 6 months)
* Cognitive impairment limiting ability to understand instructions during orientation
* Other conditions known to influence bone health or body composition as determined by the investigator
* Patients at risk for cardiovascular disease yet have not received a routine cardiology assessment within the previous 12 months
* Bone medication (e.g. Zometa, Prolia, Forteo) use in previous 2 years

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Body Lean Mass (grams) | 12 weeks (Period 1) and 36 weeks (Period 2)
  Total body lean mass assessed by Dual Energy X-Ray Absorptiometry (DXA)
Percentage Body Fat | 12 weeks (Period 1) and 36 weeks (Period 2)
  Percentage body fat assessed by Dual Energy X-Ray Absorptiometry (DXA)

SECONDARY OUTCOMES:
6 minute walk test (6MWT) | 12 weeks (Period 1) and 36 weeks (Period 2)
  Distanced walked during a 6MWT
Vertical Jump | 12 weeks (Period 1) and 36 weeks (Period 2)
  Vertical jump from a standing height (cm)
Bone Mineral Density (BMD) | 36 weeks (Period 2)
  Bone mineral density at the spine, left hip, left distal radius and whole body as assessed by Dual Energy X-Ray Absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Fung, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of California, San Francisco, Oakland, California

IPD SHARING:
Plan to Share IPD: No